CLINICAL TRIAL: NCT04557436
Title: Phase 1, Open Label Study of CRISPR-CAR Genome Edited T Cells (PBLTT52CAR19) in Relapsed /Refractory B Cell Acute Lymphoblastic Leukaemia
Brief Title: TT52CAR19 Therapy for B-cell Acute Lymphoblastic Leukaemia (B-ALL)
Acronym: PBLTT52CAR19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18IC07
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: B Acute Lymphoblastic Leukemia
Keywords: relapsed; refractory
MeSH Terms: conditions — Burkitt Lymphoma; Recurrence

STUDY DESIGN:
Intervention Model Description: This is an open label, single-centre, phase I, cohort study using genome edited T cells to bring patients with relapsed or refractory B-cell acute lymphoblastic leukaemia (B-ALL) into remission in anticipation of a haematopoietic stem cell transplant (HSCT) that will hopefully prevent the leukaemia from returning. It involves a single infusion of allogenic T cells transduced with a self-inactivating (SIN) lentiviral vector in up to 10 subjects aged from 6 months to 18 years. The primary objective in this study is to test the safety and secondary objective will test the efficacy of this gene therapy procedure in this population.
  Patients will be enrolled following diagnosis and referral to GOSH, and will receive TT52CAR19 cells at GOSH after lymphodepleting conditioning. They will be followed on this protocol for 12 months post IMP infusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard of care (Other): Follow-up period:
  For patients achieving molecular remission by day 28, allo-HSCT will be scheduled as soon as practicable. Routine transplant care for 24 months will incorporate the disease monitoring and recording of adverse events of special interest and document elimination of PBLTT52CAR19 through the transplant conditioning period.
  For patients with refractory disease at Day 56, the monitoring of adverse events of special interest, the disease outcome will be monitored monthly up to 24 months or until a palliative therapy approach is adopted.
  Assessments will be carried out after the treatment period at the following time points: 1m, 2m, 3m, 6m, and 12m, 24m
  * Physical examination, ECOG
  * Laboratory tests
  * Vital signs (temperature, BP, HR, respiratory rate, weight)
  * Persistence of PBLTT52CAR19, VCN by qPCR in blood and bone marrow (if sampled)
  * Chimerism and MRD in blood and bone marrow (if sampled)
  * Adverse events
  * Concomitant treatments
  Interventions: Drug: PBLTT52CAR19

INTERVENTIONS:
Drug: PBLTT52CAR19 — gene therapy

SUMMARY:
PBLTT52CAR19 modified T cells are allogenic engineered human T cells (defined as TT52CAR19 +TCRαβ-) prepared for the treatment of CD19+ B cell leukaemia. The cells are from healthy adult volunteer donors and are not HLA-matched. They have been transduced to express and anti-CD19 chimeric antigen receptor (CAR19) using a lentiviral vector that also incorporates CRISPR guides for genome editing of CD52 and TRAC loci in the presence of transiently provided Cas9.

Recognition by TT52CAR19 T cells mediates eradication of CD19+ leukaemia and other CD19+ B cells through T cell mediated cytotoxicity.

This study aims to apply PBLTT52CAR19 T cells to secure molecular remission in children with relapsed/refractory B-ALL ahead of programmed allogeneic stem cell transplantation. The cells are to be used in a time-limited manner for their anti-leukaemia effects and then depleted by standard pre- transplant conditioning.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed (second or subsequent bone marrow relapse or bone marrow relapse after allo-SCT) or refractory (not achieving an initial complete response (CR) after 2 cycles of standard chemotherapy) CD19-positive B-acute lymphoblastic leukaemia
* Morphologically confirmed with leukemic blasts in the bone marrow or a quantifiable MRD load of 1x10-4 (by multiparameter flow cytometry and/or quantitative polymerase chain reaction)
* Eligible and fit for allogeneic hematopoietic stem cells transplantation with suitable donor available
* Estimated life expectancy ≥ 12 weeks
* Lansky (age < 16 years at the time of assent/consent) or Karnofsky (age ≥ 16 years at the time of assent/consent) performance status ≥ 50 Eastern Cooperative Oncology Group ECOG performance status < 2

Exclusion Criteria:

* Patients/parents unwilling to undergo a follow-up for 15 years
* Foreseeable poor compliance to the study procedures
* CD19-negative B-cell leukaemia
* Evidence of disease progression after cytoreduction
* Uncontrollable CNS leukaemia or neurological symptoms defined as CNS grade 3 (per National Comprehensive Cancer National guidelines). Patients developing grade 3 CNS disease at any time after enrolment will be excluded.
* Absence of suitable HLA matched or mismatched donor
* Weight < 6 kgs
* Presence of donor-specific anti-HLA antibodies directed against PBLTT52CAR19
* GvHD requiring systemic therapy
* Systemic steroid therapy prednisolone >0.5mg/kg/day
* Known hypersensitivity to any of the test materials or related compounds
* Active bacterial, fungal, or viral infection not controlled by a standard of care anti-microbial or anti-viral treatment. Uncontrolled bacteraemia/ fungaemia is defined as the ongoing detection of bacteria/fungus on blood cultures despite antibiotic or anti-fungal therapy.
* Uncontrolled viraemia is defined as rising viral loads on two consecutive occasions despite antiviral therapy.
* Risk of pregnancy or non-compliance with contraception (if applicable). Girls of childbearing potential must have been tested negative in a pregnancy test within 14 days prior to inclusion.
* Lactating female participants unwilling to stop breastfeeding
* Intrathecal methotrexate within 4 weeks or intrathecal chemotherapy (e.g Ara-C) within 2 weeks of lymphodepletion
* Less than 2 half-lives from prior therapy with immune checkpoint pathway modifiers to lymphodepletion
* Prior CAR19 therapy known to be associated with ≥Grade 3 cytokine release syndrome (CRS) or ≥Grade 3 drug-related CNS toxicity

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
B-ALL remission | 28 days
  The main benefit expected from PBLTT52CAR19 for anti-CD19 activity leading to anti-leukemic effect and induction of remission in children with refractory/relapsed B-ALL. Patients who achieve molecular remission will become eligible to receive an allo-HSCT that would otherwise be considered futile.Remission of B-cell acute lymphoblastic leukaemia (B-ALL) in anticipation of a haematopoietic stem cell transplant (HSCT that would otherwise be considered futile.

CONTACTS AND LOCATIONS:
Overall Officials: Waseem Qasim, Prof, Principal Investigator — UCL GOSH Institute of Child Health; Paul Veys, PhD, MD, Study Director — Great Ormond Street Hospital; Kanchan Rao, PhD, MD, Study Director — Great Ormond Street Hospital; Ajay Vora, Prof, MD, Study Director — Great Ormond Street Hospital
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ottaviano G, Georgiadis C, Gkazi SA, Syed F, Zhan H, Etuk A, Preece R, Chu J, Kubat A, Adams S, Veys P, Vora A, Rao K, Qasim W; TT52 CRISPR-CAR group. Phase 1 clinical trial of CRISPR-engineered CAR19 universal T cells for treatment of children with refractory B cell leukemia. Sci Transl Med. 2022 Oct 26;14(668):eabq3010. doi: 10.1126/scitranslmed.abq3010. Epub 2022 Oct 26. PMID 36288281